CLINICAL TRIAL: NCT04270656
Title: Liver and Metabolic Effects of Insulin Pump Therapy in a Population of Type 2 Diabetics with Non-alcoholic Hepatic Steatosis
Brief Title: Liver and Metabolic Effects of Insulin Pump Therapy in Diabetics Type 2 with Non-alcoholic Hepatic Steatosis
Acronym: STEATO-POMPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC19_0449
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin pump therapy (Experimental)
  Interventions: Procedure: Insulin pump therapy
- Multi-injection treatment ( MDI ). (Active Comparator)
  Interventions: Procedure: Multi-injection treatment ( MDI ).

INTERVENTIONS:
Procedure: Insulin pump therapy — 5-day hospitalization in case of randomization in the insulin pump group (insulin pump establishing in according to the recommendations of the HAS)
  Arms: Insulin pump therapy
Procedure: Multi-injection treatment ( MDI ). — Corresponds to an outpatient visit if the patient is randomized into the multi-injection group
  Arms: Multi-injection treatment ( MDI ).

SUMMARY:
The prevalence of fatty liver disease (NAFLD: Non-Alcoholic Fatty Liver Disease or to a more severe degree NASH: Non-Alcoholic SteatoHepatitis) reached 40-70% in subjects with type 2 diabetes (T2D). NAFLD can be easily detected by performing a hepatic ultrasonography. The presence of a NAFLD is positively correlated with the severity of insulin resistance and dysglycemia in this population. The presence of NAFLD worsens the prognosis of T2D with an increased cardiovascular risk. This hepatic impairment would also increase the risk of microvascular complications, especially nephropathy. Conversely, T2D increases the risk of transition from NAFLD to NASH and then to hepatic fibrosis and its related complications (cirrhosis, hepatocellular carcinoma). The risk of progression of liver steatosis to fibrosis is also more important as diabetes and insulin resistance are more severe.

In addition to diabetes and insulin resistance, other risk factors are associated with more severe liver damage such as changes in microbiota. Indeed, it has already been described a smaller amount of bacteroides in the microbiota of subjects with T2D and the most severe hepatic impairment. The treatment of NAFLD/NASH is poorly codified without approved drugs in this indication, while many phase 3 trials with candidate drugs are undergoing. Life-style measures (physical activity and low carbohydrate/calorie diet) can limit the progression from NAFLD to more severe liver fibrosis. Some bariatric surgery studies have also shown good results in this situation. Pharmacological interventions are also reported with proven efficacy of pioglitazone, vitamin E and orlistat.

The OPT2MISE study has recently shown the superiority of insulin pump (or continuous sub-cutaneous insulin infusion: CSII) compared to multiple daily insulin injections (MDI) to improve glycemic control in a population of patients with T2D in failure of well-titrated MDI. In addition, treatment with CSII showed a 45% decrease in insulin resistance (assessed by HOMA-IR) in a population of newly diagnosed T2D.

In light of these data, investigators hypothesize that the introduction of insulin pump treatment in a population of subjects with T2D and NAFLD, by improving insulin sensitivity, could reduce fatty liver content compared to standard MDI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male / female 35/70 years (including ranges) with T2D ≥ 1 year
* Benefiting from the indication of use of the free Freestyle glucose meter
* Treatment with multi-injection insulin therapy comprising a daily injection of basal insulin (Glargine U100, Glargine U300, Degludec) and at least 2 daily injections of an insulin analogue (lispro, aspart or glulisine) +/- metformin, dipeptidyl peptidase-4 (DPP4) and/or sodium-glucose cotransporter type 2 (SGLT2) at a dose stable for at least 3 months.
* For women of childbearing age, oestro-progestative pill, IUD, implant.
* 11% ≥ HbA1c ≥ 6.5%
* Presence of hepatic steatosis according to the ultrasonography
* Absence of chronic alcoholic intoxication
* Absence of chronic viral hepatitis or other chronic liver diseases (eg hemochromatosis ...)

Exclusion Criteria:

* Type 1 diabetes
* Contraindication to pump treatment
* Treatment with anti-diabetics or other than metformin, dipeptidyl peptidase-4 (DPP4) and/or sodium-glucose cotransporter type 2 (SGLT2)
* Treatment with basal inulin of Levemir
* Contraindication to performing MRI
* Chronic alcohol abuse (after alcohol consumption> 20g / day in men and> 10g / day in women) according to the medical examination
* Chronic viral hepatitis based on HBV and HCV serology results
* Hemochromatosis according to the martial assessment
* Other toxic or drug hepatitis
* Severe hepatic pathology: hepatic cirrhosis, hepatocellular carcinoma
* Severe renal insufficiency (MDRD <30 ml / min)
* Severe and progressive cardiovascular pathology
* Treatment (permanent or intermittent) with glucocorticoids
* Treatment known to improve hepatic steatosis (glitazone, vitamin E, orlistat)
* history or bariatric surgery project for the duration of the study
* Drug treatment likely to cause hepatic steatosis (amiodarone, carbamazepine, tamoxifen, valproate, clozapine, anti-retroviral drugs) unless the dose has been stable for ≥ 3 months
* Guardianship, curatorship or safeguard of justice

Ages: 37 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Variation of hepatic steatosis, between the insulin pump therapy (CSII) vs Multi injection treatement (MDI) groups. | 6 months
  Change of fatty liver by MRI quantification

SECONDARY OUTCOMES:
In the CSII group : avantage of an insulin pump treatment on the fatty liver between inclusion and the 6th month, | 6 months
  Variation of hepatic steatosis (MRI quantization by gradient echo sequences & centralized reading
In the CSII group : avantage of an insulin pump treatment on the fatty liver (quantified by MRI), between inclusion and the 12th month, | 12 months
  Variation of hepatic steatosis (MRI quantization by gradient echo sequences & centralized reading
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months, on hepatic biological parameters and non-invasive biomarkers of fatty liver (FLI) and of fibrosis of the liver (FIB-4 and NAFLD Score), | 6 months
  Liver fonction (AST ; ALAT ; GGT ; PAL ; Ferritin) Test-fibrosis score criteria (FIB- 4 and NAFLD Score) ; FLI
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on insulin sensitivity | 6 months
  dosage of plasma adiponectin
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on insulin sensitivity | 6 months
  calculation of the modified HOMA-IR index (peptide C, blood sugar),
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on glycemic balance | 6 months
  HbA1c dosages
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on the total daily insulin dose | 6 months
  daily insulin dose record
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on lipid profile • the inflammatory condition | 6 months
  total cholesterol
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on lipid profile • the inflammatory condition | 6 months
  LDL-cholesterol
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on lipid profile • the inflammatory condition | 6 months
  HDL-cholesterol
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on lipid profile • the inflammatory condition | 6 months
  triglycerides (TG)
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on lipid profile • the inflammatory condition | 6 months
  fatty-free acids
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on lipid profile • the inflammatory condition | 6 months
  ApoB,
Evaluate the effectiveness of a CSII vs MDI treatment, between randomization and 6 months on CRPus | 6 months
  Ultra-sensitive C-reactive protein (CRPus)
Evaluation of quality of life | 6 months
  DTSQ
Evaluation of quality of life | 6 months
  SF36
Safety analysis at 6 months: comparison the first 6 months, in the CSII and MDI groups: | 6 months
  Reporting by patient of all severe hypoglycemia during the study
Safety analysis at 6 months: comparison the first 6 months, in the CSII and MDI groups: | 6 months
  Reporting by the patient of all episode of ketoacidosis during the study
Calculation of the sensitivity values of the FLI for the detection of fatty liver in this population, | 6 months
  quantification of hepatic MRI as Gold Standard.
Calculation of the specificity values of the FLI for the detection of fatty liver in this population, by using the quantification of hepatic MRI as Gold Standard. | 6 months
  quantification of hepatic MRI as Gold Standard.
Calculation of the positive predictive values of the FLI for the detection of fatty liver in this population, by using the quantification of hepatic MRI as Gold Standard. | 6 months
  quantification of hepatic MRI as Gold Standard.
Calculation negative predictive values of the FLI for the detection of fatty liver in this population, by using the quantification of hepatic MRI as Gold Standard. | 6 months
  quantification of hepatic MRI as Gold Standard.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU, Angers
  - CHU, Caen
  - CHU, Dijon
  - CHU, La Rochette
  - Hospices Civils, Lyon
  - Nantes UH, Nantes
  - CHU, Poitiers
  - CHU de Rennes, Rennes
  - CHU, Toulouse

IPD SHARING:
Plan to Share IPD: No